CLINICAL TRIAL: NCT04785079
Title: Qualification of Instrument Assisted Soft Tissue Mobilization Induced Hyperemia Using Musculoskeletal Ultrasound
Brief Title: Instrument Assisted Soft Tissue Mobilization Effect on Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Collaborators: Thomas Zeller (Unknown); Tyler Corbin (Unknown); Alyssa Nieves (Unknown)
Responsible Party: Principal Investigator, Dr. Rob Sillevis,, Assistent Professor, Florida Gulf Coast University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-34
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Asymptomatic Condition
Keywords: Instrument assisted soft tissue mobilization; Musculoskeletal Ultrasound Imaging; Bood circulation; Perception
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study using a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Graston effect medial arch, plantar fascia, and trapezius (Experimental): Pre and post Graston change in blood flow at the medial arch foot, plantar fascia, and the trapezius region
  Interventions: Procedure: Graston Instrument assisted Soft tissue Mobilization

INTERVENTIONS:
Procedure: Graston Instrument assisted Soft tissue Mobilization — Instrument assisted soft tissue mobilization using the Graston tool and technique for 3 minutes on each of the three locations

SUMMARY:
This study is designed to evaluate the short term change in blood flow in the superficial human tissue layers after the application of 3 min Graston instrumented assisted soft tissue mobilization on the plantar aspect of the foot and the trapezius muscle.

DETAILED DESCRIPTION:
Instrument assisted soft tissue mobilization (IASTM) is a commonly used physical therapy intervention. Graston ® technique is a form of IASTM that requires completion of a certification course and utilizes specific stainless-steel tools. IASTM has been found to improve range of motion, pain and patient reported function in pathological individuals. One method by which these improvements are thought to occur is by increasing blood flow. Increased blood flow brings nutrients and oxygen to the area and is thought to contribute to tissue remodeling. There is very limited research investigating blood flow changes following IASTM. In order to measure blood flow changes following IASTM, doppler ultrasound may be used. There are no studies to our knowledge quantifying changes in blood flow following IASTM using ultrasound. Power doppler approximates perfusion by detecting a frequency shift from movement of red blood cells and color is then encoded proportionally to the number of red blood cells. Power doppler imaging quantification (PDIQ) is a feature of musculoskeletal ultrasound (MSK) that compares the number of color pixels and the intensity of color within these pixels to grey scale pixels within a given image. The aim of this study is to determine if there is an increase in blood flow in the trapezius, plantar fascia and medial arch of the foot measured following IASTM. Blood flow was measured by using PDIQ ratio in the doppler setting of MSK ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* A-symptomatic individuals over the age of 18

Exclusion Criteria:

* Anyone under 18 and anyone with any conditions contraindicated for IASTM including compromised tissue integrity, deep vein thrombosis (DVT), area of infection in the treatment area, or acute fracture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
GE LOGIQe ultrasound machine to measure maximum power doppler imaging quantification (PDIQ) ratios | One day measure-First measure will be taken before the treatment intervention, immediate after the intervention and three minutes afterward. Total time for the experiment is 15 minutes
  ultrasound images are used to calculate the ratio of color to grey scale pixels called the power doppler quantification ratio (PDIQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Gulf Coast University, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No